CLINICAL TRIAL: NCT05082220
Title: Comparison of the Spread Level During Thoracic Erector Spinae Plane Block Using Two Volumes of Local Anesthetics
Brief Title: Analysis of Spread Level During Thoracic Erector Spinae Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dongsan Hospital
Record Dates: First submitted 2021-09-30; First posted 2021-10-18 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Pain; Radiculopathy, Cervical
MeSH Terms: conditions — Pain; Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 ml ESPB group (Experimental): ESPB group using 10 ml mixture of local anesthetics and contrast medium using ultrasound and fluoroscopy
  Interventions: Procedure: Erector spinae plane block
- 20 ml ESPB group (Experimental): ESPB group using 20 ml mixture of local anesthetics and contrast medium using ultrasound and fluoroscopy
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — fascial plane injection using ultrasound and fluoroscopic guidance

SUMMARY:
The primary purpose of this study was to identify the ESPB spread level in the craniocaudal direction when performed at the T2 level. The secondary purpose was to determine the incidence of spread into epidural, paravertebral, intercostal, and intravascular injections with ESPB

DETAILED DESCRIPTION:
The ESPB requires ultrasound guidance which enables visible local anesthetic spread underneath the erector spinae muscles. The spinalis, longissimus thoracis, and iliocostalis muscles comprise the ES muscles, which run vertically along both sides of the vertebral column from the sacrum up to the skull base. The ESPB can be performed in the cervical, thoracic, and lumbar regions. Among them, upper or mid thoracic ESPB has been used more widely compared to cervical and lumbar regions. Previous cadaveric studies on the ESPB at the T5 level using computed tomography (CT) reconstruction or direct dissection demonstrated the extensive craniocaudal distribution of methylene blue ranging from T1 to T8 vertebral segments deep to the ES muscles and variable involvement of epidural, paravertebral, and intercostal spaces. The ESPB performed at the T2 level of the cadaver demonstrated an injected dye distribution ranging from C4 to T10. Also, 36% of cadavers showed the spread of an injected dye to the ventral, dorsal ramus, paravertebral space, and even the contralateral side. The exact mechanism of action of ESPB remains unclear. A recent study suggested that the analgesic effect of ESPB could be obtained by blocking the ventral and dorsal ramus of the spinal nerves by passing through the costotransverse foramen. However, in clinical practice, we can encounter highly variable clinical outcomes or sensory block after the ESPB. The study of the physical spread of the injected agent can be used to predict the clinical result and elucidate the possible mechanism of action of ESPB.

ELIGIBILITY:
Inclusion Criteria:

* cervical facet joint arthrosis
* cervical foraminal stenosis
* cervical herniated intervertebral disc
* myofascial pain syndrome of upper back muscle

Exclusion Criteria:

* allergy to local anesthetics or contrast medium
* pregnancy
* prior history of cervical spine surgery
* coagulation abnormality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
spread level in the cranio-caudal direction | Baseline, 5 minutes after erector spinae plane block
  fluoroscopic contrast medium spread level in the cranio-caudal direction

SECONDARY OUTCOMES:
Number of participant showing epidural spread | baseline, 5 minute after erector spinae plane block
  Number of participant showing epidural spread by analysis of fluoroscopic image
Number of participant showing intercostal spread | baseline, 5 minute after erector spinae plane block
  Number of participant showing intercostal spread by analysis of fluoroscopic image
Number of participant showing paravertebral spread | baseline, 5 minute after erector spinae plane block
  Number of participant showing paravertebral spread by analysis of fluorosocpic image
Number of participant showing intravascular spread | baseline, 5 minute after erector spinae plane block
  Number of participants showing intravascular spread by analysis of fluoroscopic image

CONTACTS AND LOCATIONS:
Overall Officials: Ji H Hong, Principal Investigator — Keimyung University
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided